CLINICAL TRIAL: NCT04670510
Title: Aerobic Exercise for Optimizing Cognitive and Brain Health in Remitted Late-Life Depression
Brief Title: Fitness for Brain Optimization for Late-Life Depression
Acronym: FIT BOLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Swathi Gujral, Assistant Professor of the Department of Psychiatry at the University of Pittsburgh, School of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY20080088; K23MH125074 (NIH)
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Depression in Old Age
Keywords: Depression; Exercise; Late-Life; Cognitive Impairment; Brain Health
MeSH Terms: conditions — Depression; Motor Activity; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise (Experimental): The Aerobic Exercise (AE) condition will involve 150-minutes of moderate-intensity AE per week for 6-months and will involve a graded decline in supervision. Supervised AE will occur in groups, though each participant's AE prescription will be personalized based on baseline exercise capacity, as assessed by a maximal cardiopulmonary fitness test. Supervised AE sessions will involve the treadmill, elliptical, and/or bike, and routines will be varied to promote adherence. Supervised AE sessions will gradually increase to 50-minutes per session; however, participants will be encouraged to engage in home-based AE sessions according to their own preference of length and frequency in order to achieve 150 minutes of AE per week.
  Interventions: Other: On-site AE; Other: At-home AE
- Social Engagement (Active Comparator): The Social Engagement (SE) condition will be designed to control for the social component of the AE intervention (i.e., supervised on-site sessions with professional staff, frequent phone contact from study staff). A variety of enjoyable group-based activities centered around the dimensions of wellness (spiritual wellness, physical wellness, emotional wellness, etc.) will be scheduled throughout the intervention. This condition will involve once weekly meetings (grand total of ~26 sessions). Some participants will meet in-person and others will meet remotely via zoom (this will vary week to week) to increase flexibility to accommodate participant availability to attend as many sessions as possible.
  Interventions: Other: Social Engagement (SE)

INTERVENTIONS:
Other: On-site AE — Participants will attend on-site supervised AE sessions 3 times per week for the first 6 weeks, twice weekly for weeks 7-12; once weekly for weeks 13-18.
  All supervised sessions will start and end with 5-minute warm-up and cool-down and will involve exercise on the treadmill, elliptical, and/or bike. During AE sessions, participants will exercise so that their heart rate is approximately 65% of their peak heart rate and gradually increase the intensity of exercise so that their heart rate is between 70 and 85% of their peak heart rate. All participants will wear heart rate monitors and encouraged to exercise in their target heart rate zone. Supervised AE sessions will gradually increase to 50-minutes per session
  Arms: Aerobic Exercise
Other: At-home AE — Participants will increase at-home AE during the 6-month intervention period with weeks 19-26 occurring entirely at-home. As participants transition to home-based exercise, they will be equipped with a polar heart rate monitor and will be instructed to use this to record average heart rate during each exercise session. On a log sheet, they will record both average heart rate during exercise and average subjective rating of perceived exertion (RPE) during each exercise session.
  Arms: Aerobic Exercise
Other: Social Engagement (SE) — To control for the social component of the AE intervention participants in the SE group will be invited to attend at total of 25 group meetings over the course of the 6-month study period.
  Arms: Social Engagement

SUMMARY:
Cognitive impairment and brain abnormalities are common and persist after depression remission in those with Late Life Depression (LLD), compounding dementia risk in both individuals with acute and remitted LLD (rLLD). In this study, investigators will examine systemic neural and cognitive benefits of aerobic exercise training in older adults with remitted LLD. This will generate preliminary data regarding neural targets of aerobic exercise training that may translate to cognitive benefits in those with rLLD, a population who remains at high risk for dementia despite successful treatment of depression.

DETAILED DESCRIPTION:
Significance:

The population of adults aged >65 years in United States is expected to nearly double between 2012 and 2050, with a projected estimate of 83.7 million adults aged >65 years by 2050. The prevalence of depressive symptoms among older adults ranges 15 - 27% in the community and up to 37% in primary care settings. Though subclinical depressive symptoms are more prevalent than Major Depression (MDD) among older adults (MDD: 5.5% prevalence), rates of MDD in older people have been rising over the past two decades. Late-life depression (LLD) results in enormous economic, public health, and caregiver burden. This high economic cost consists of both direct and indirect costs (e.g., increased use of medical resources, need for unpaid family caregiving). Further, LLD exacerbates chronic medical illness burden and confers the greatest risk for mortality across all mental health conditions in aging. LLD also increases disability risk, with one report estimating 79% of LLD having functional limitations. Importantly, those with LLD are at a twofold increased risk for dementia relative to the general aging population, which has catastrophic implications for the long-term economic and public health burden of LLD.

Background:

Older adults with LLD are particularly predisposed to accelerated rates of cognitive decline and progression to dementia. While nearly half of those with LLD have significant cognitive impairment, cognitive deficits are inadequately addressed using conventional antidepressant treatments. Exercise has emerged as the leading non-pharmacological approach to improve cognition and reduce dementia risk in aging. AE interventions in older adults, over as short as 6-months, have been shown to improve performance in cognitive functions (i.e., executive function) and brain regions and networks (i.e., PFC, HC, DMN) that are most sensitive to the neurotoxic effects of LLD. However, our knowledge of AE-related cognitive and brain changes in aging are primarily drawn from AE trials conducted in populations at low risk for dementia. Though an emerging literature supports the benefits of AE for cognitive and brain health in those with MCI, these studies systemically exclude psychiatric populations. By excluding those with LLD, existing studies are overlooking a subsample of older adults at ultra-high risk for dementia for whom the cognitive and neural benefits of AE training may be particularly consequential. This necessitates a better understanding of the potential of AE training to target systemic brain features and cognition in those who have had LLD.

Impact:

This study will probe whether AE -related systemic brain changes may be mechanistic targets for improving cognition in those with rLLD. It cannot be assumed that AE effects on brain health will be consistent across populations with varying levels of brain-related abnormalities. This study allows for an initial exploration of the extent to which AE effects on cognitive and brain health in those with rLLD are similar to and distinct from AE effects on cognitive and brain health in older adults who 1) are cognitively normal or 2) do not have a history of LLD, for whom the majority of the AE brain health and cognition literature is based.

Study Aims:

Aim 1. Examine AE effects on structural and functional neuroimaging markers of brain health in rLLD. H1a. AE relative to SE will result in greater preservation of gray matter integrity in areas shown to be abnormal in LLD (HC and PFC) but not in the occipital cortex or thalamus. H1b. AE relative to SE will result in enhanced functional connectivity within the DMN and cross-network connectivity between the DMN and ECN. H1a. Separate ANCOVA models will be used to examine intervention group differences in change in HC and thalamus volume (mm3) and cortical thickness of PFC regions (i.e., dorsolateral PFC, medial orbitofrontal cortex, and ACC) and the occipital cortex, from baseline to 6-months, all of which will be estimated using semiautomated segmentation methods. H1b. Primary analysis of resting state functional magnetic resonance (fMRI) data will involve ANCOVAs to examine group differences in change in within-network DMN connectivity and cross-network DMN-ECN connectivity using summary network connectivity measures. Linear mixed models testing group x time interaction effect for PCC-whole brain voxel-wise connectivity maps will be used in secondary analyses.

Aim 2. Examine AE effects on cognitive functioning in rLLD. H2. AE relative to SE will improve cognitive performance, showing the greatest effect for executive functioning. Primary analyses will use ANCOVA models to examine group differences in change in performance for each cognitive domain from baseline to 6-months. Secondary analyses will involve random slopes and random intercept models for repeated longitudinal data to examine group differences in trajectory of change in performance for each cognitive domain over 6-months across three timepoints (baseline, 3-months, 6-months). Exploratory analyses will also involve a comparison of group differences in trajectory of change in objective cognitive performance relative to subjective reports of cognitive functioning.

(Exploratory) Aim 3. Explore the extent to which AE-related structural and functional brain changes are associated with AE-related cognitive changes in those with rLLD. H3. AE-related changes in HC and/or PFC integrity and/or DMN connectivity will be associated with AE-related cognitive changes. H3. Pearson's correlations will be used to examine the association between change in brain outcomes showing an effect of AE training and change in performance for cognitive domains showing an effect of AE training.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 60+ years
2. Major Depressive Episode in older adulthood (since age 55)
3. Current level of depressive symptoms does not meet criteria for a Major Depressive Episode
4. Ambulatory without pain or the assistance of walking devices
5. Able to speak and read English
6. Exercise level of <100 minutes per week on average
7. Medical clearance by primary care physician (PCP)
8. Living in community for duration of the study
9. Reliable means of transportation
10. No diagnosis of a neurological disease
11. Eligible to undergo MRI

Exclusion Criteria:

1. Current diagnosis of a Major Depressive Episode
2. Psychosis
3. Significant suicide risk (i.e., current, active suicidal ideation with a plan)
4. Electroconvulsive therapy within the past 12 months
5. Engaging in moderate-intensity exercise >100 minutes per week on average
6. Current treatment for cancer - except non-melanoma skin
7. Neurological condition (MS, Parkinson's, Dementia, MCI) or brain injury (Stroke)
8. Substance Use disorder in the past 3-months
9. Current treatment for congestive heart failure, angina, uncontrolled arrhythmia, deep vein thromboses (DVT) or other cardiovascular event
10. Myocardial infarction, coronary artery bypass grafting, angioplasty or other cardiac condition in the past year including uncontrolled hypertension
11. Regular use of an assisted walking device
12. Presence of metal implants (pacemaker, stents) that would be MR ineligible
13. Claustrophobia
14. Color Blindness
15. Significant visual or hearing impairments that would preclude neuropsychological assessment or communication with study staff via a virtual format (videoteleconference)
16. Not fluent in English
17. Not medically cleared by PCP
18. Traveling consecutively for 3+ weeks during the study
19. MOCA (<20 to exclude) and MADRS (>9 to exclude)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Cardiovascular Fitness at 6 months | Baseline and 6-months
  Cardiorespiratory fitness will be measured via a cardiopulmonary exercise test (CPET) indicated by maximal VO2 on a motorized treadmill. while measuring oxygen utilization via Parvo Medics True one metabolic cart. The test follows a modified Balke protocol in which speed remains constant with the intensity being increased every two minutes via a raise of 2.0% of the incline. The speed was an agreed upon speed between participant and staff (between 2.0 and 4.0 mph). The test will conclude when the participant reaches 85% of age predicted maximal heart rate, rating of perceived exertion (RPE) equal to or greater than 15 for those who have blunted heart rate response due to beta block medication, or volitional termination by participant.
Changes from baseline in Brain Structure and Function at 6 months | Baseline and 6-months
  Brain imaging conducted with a 7 Tesla scanner. Of particular interest are changes in hippocampal volume. This measurement is reported in mm^3, with higher numbers indicating higher levels of gray matter in the hippocampal region. Changes in prefrontal cortical thickness are also of interest, measured in mm. Brain functional network changes of interest are changes in intra- and inter-connectivity of the default-mode and executive control large-scale brain networks.
Changes from baseline in depressive symptoms at 6 months | Baseline and 6-months
  Given that all participants will have a recent history of depression, and may have lingering low level symptoms or may even relapse, depressive symptoms will be assessed using the Montgomery Asberg Depression Rating Scale (MADR; score ranges from 0 [better] to 60 [worse]), a clinician administered measure of depression severity.
Depressive Symptoms | Continuously up to every 6-weeks for 6 months
  For the frequent assessment of depressive symptoms during the intervention while minimizing participant and clinician burden, the Patient Health Questionnaire-9 item version (PHQ-9; score ranges from 0 [better] to 27 [worse]), a self-report questionnaire, will be administered.
Change from baseline in Cognitive Function at 6 months | Baseline and 6-months
  Assessed with a comprehensive Neuropsychological Battery. The primary cognitive outcome will be assessed using a composite score (mean) of standardized scores (Z-scores) from the following executive functioning tests from the NIH toolbox: 1) Dimensional Change Card Sort Test (set-shifting), Flanker Inhibitory Control and Attention Test (inhibition), List Sorting Working Memory Test (working memory).

SECONDARY OUTCOMES:
During-intervention physical activity levels | Continuously up to every 2 months for 6 months
  Participants will wear wrist Actigraphy to monitor physical activity levels
Change from baseline in amount of physical activity at 6 months | Baseline and 6-months
  Participants will wear wrist Actigraphy to monitor amount of physical activity
Changes from baseline in intensity of physical activity at 6 months | Baseline and 6-months
  Participants will wear wrist Actigraphy to monitor intensity of physical activity
Change from baseline in Subjective Cognitive Function at 6 months | Baseline and 6-months
  Subjective reports of cognitive functioning will also be assessed using the Measurement of Everyday Cognition (E-Cog; scores range from 1 [better] to 4 [worse]), given that those with a recent history of LLD may be likely to underestimate their cognitive abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Swathi Gujral, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Western Psychiatric Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Current and future investigators, both internal and external, may have access to de-identified data; however only group data would be shared.

DOCUMENTS (1):
  • Informed Consent Form (2024-08-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT04670510/ICF_000.pdf